CLINICAL TRIAL: NCT04036942
Title: Ablation Of The Esophagogastric Junction With Hybrid Argon Plasma Vs Mucosectomy With Band in Patients With Gastroesophageal Reflux Disease Without Hiatal Hernia
Brief Title: Antireflux Ablation Therapy (ARAT) Vs Antireflux Mucosectomy (ARMS) In The Management Of Gastroesophageal Reflux Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: problems with participants enrollment
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-2019-3601-179
Record Dates: First submitted 2019-07-25; First posted 2019-07-30 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastroesophageal Reflux Disease (GERD); ARAT; ARMS
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: A simple randomized, comparative (pretreatment and posttreatment), prospective clinical trial will be carried out among the group of patients managed with ARAT and ARMS
Who Masked: Investigator
Masking Description: The investigator in charge of capturing the data will only know if the patients received an A or B treatment without knowing the meaning of these letters; the endoscopist who carries out the procedure and the patient will be aware that group A corresponds to management with ARAT and group B to management with ARMS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hybrid argon plasma. (Active Comparator): After diagnostic endoscopy investigators will proceed to use argon plasma probe for marking 270 grades around the esophagogastric junction preserving part of the mucosa towards the greater curvature, then investigators will use the jet included in the argon plasma probe with effect 20 to 40 system for the injection of the background submucosa in the marking area, applying 0.9% saline solution with methylene blue, to achieve adequate Submucosal elevation for application or argon plasma with high voltages (100 watts, 1.5 liters / min) using forced coagulation mode, applying plasma argon to 1cm above the Z line in the esophageal mucosa and 2cm below it towards the gastric mucosa, argon will be applied until a "carbonization" effect of the mucosa is achieved, once the application of the therapy is performed mucosal lavage and immersion technique to corroborate integrity and continuity of the gastrointestinal tract and rule out immediate complications
  Interventions: Procedure: Ablation of the gastroesophageal junction with hybrid argon plasma
- Band mucosectomy (Active Comparator): After diagnostic endoscopy investigators will proceed to use the tip of a polypectomy snare for marking 270 grades around the esophagogastric junction preserving part of the mucosa towards the greater curvature, then investigators will perform submucosal elevation with the injection of 0.9% saline with carmine indigo and adrenaline 1:10000, after adequate submucosal elevation investigators will proceed with the help of a band ligation cap to suction and release the elastic band in the previously marked and elevated tissue, proceeding to resect the previously ligated tissue with polypectomy loop below the elastic band with forced coagulation (Effect 2, 40 W), until the marked mucosa is completely resected (average used of 5 elastic bands, reviewing the work area for complications like bleeding or perforation.
  Interventions: Procedure: mucosectomy with band of the gastroesophageal junction

INTERVENTIONS:
Procedure: Ablation of the gastroesophageal junction with hybrid argon plasma — In the management group with argon plasma hybrid after marking 270 degrees of the esophagogastric junction, submucosal elevation and argon plasma burn of the marked and elevated area is performed.
  Other Names: ARAT
  Arms: Hybrid argon plasma.
Procedure: mucosectomy with band of the gastroesophageal junction — In the management group with mucosectomy after marking 270 degrees of the esophagogastric junction, a submucosal elevation of the marked area is performed to subsequently perform ligation and resection with a hot snare below the ligation area.
  Other Names: ARMS
  Arms: Band mucosectomy

SUMMARY:
Gastroesophageal reflux disease has a high global prevalence, proton pump inhibitors are the cornerstone in the management but 10-20% of the patients are refractory to these, surgical treatment being an option of treatment in these patient but its associated with high morbidity, as well as a greater possibility of early therapeutic failure, for these reasons new therapies are in development being the mucosectomy with band and ablation of the esophagogastric junction with hybrid argon plasma options widely available that can offer a viable therapeutic option for patients with difficult control of symptoms or those who does not want to receive continuous medical treatment or surgical treatment. The aims of the study is to evaluate the safety and efficacy of this new techniques in the management or gastroesophageal reflux disease without hiatal hernia.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease is a disease with high global prevalence, reaching rates of 19.6 and 40% in our country, for which it is one of the most common reasons for medical care and although a clinical response is obtained in an 80-90% of patients with the use of proton pump inhibitors, the rest of the patients represents a medical challenge; surgical and endoscopic treatment being within the treatment options, the former having a high related morbidity (perforation, vagal nerve injury, postoperative dysphagia, etc), its duration is suboptimal and a second operation is associated with more surgical complications and morbidity, as well as a greater possibility of early therapeutic failure. For all these reasons, new endoluminal therapies have begun to be planned, including transoral fundoplication and radiofrequency ablation of the esophagogastric junction, these with controversial results and with the need of the use of special accessories and instruments that are not widely available; mucosectomy with band and ablation of the esophagogastric junction with hybrid argon plasma are widely available procedures in medical centers, offering a viable therapeutic option for patients with difficult control of symptoms or those who does not want to receive continuous medical treatment or surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes over 18 years and under 90 years with a diagnosis of GERD and who are under medical treatment and who do not want surgical treatment.
* Confirmed diagnosis of GERD as follows:

Positive pHmetry. Positive endoscopy (Esophagitis grade C, D, stenosis or EB)

* Esophagogastric junction Hill I-III
* Total or partial response to proton pump inhibitors
* Patient who does not wish to take medication for the treatment of gastroesophageal reflux in the long term or indefinitely or refractory GERD

Exclusion Criteria:

* Patients who do not accept the signature of the informed consent
* Postoperative fundoplication patients for GERD
* Patients with extraesophageal symptoms.
* Pregnant women.
* Patients with hiatal hernia larger than 3 cm or Hill type IV.
* Patients with major esophageal motility disorders.
* Patients with portal hypertension and presence of esophageal varices
* Patients with hemophilia or some haematological disorder that is difficult to control
* Patients with malignant pathology of the esophagus or Gastroesophageal Junction (GEJ).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
efficacy of management with ARAT and ARMS in reducing the total percent acid exposure time | 3, 6 and 12 months
  the investigators will compare the percentage of improvement in esophageal Ph metry before and after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Oscar V Hernandez Mondragon, MD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Centro Medico Nacional Siglo XXI Hospital de Especialidades, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hedberg HM, Kuchta K, Ujiki MB. First Experience with Banded Anti-reflux Mucosectomy (ARMS) for GERD: Feasibility, Safety, and Technique (with Video). J Gastrointest Surg. 2019 Jun;23(6):1274-1278. doi: 10.1007/s11605-019-04115-1. Epub 2019 Feb 7. PMID 30734179
- [Background] Gyawali CP, Kahrilas PJ, Savarino E, Zerbib F, Mion F, Smout AJPM, Vaezi M, Sifrim D, Fox MR, Vela MF, Tutuian R, Tack J, Bredenoord AJ, Pandolfino J, Roman S. Modern diagnosis of GERD: the Lyon Consensus. Gut. 2018 Jul;67(7):1351-1362. doi: 10.1136/gutjnl-2017-314722. Epub 2018 Feb 3. PMID 29437910
- [Background] Manner H, Neugebauer A, Scharpf M, Braun K, May A, Ell C, Fend F, Enderle MD. The tissue effect of argon-plasma coagulation with prior submucosal injection (Hybrid-APC) versus standard APC: A randomized ex-vivo study. United European Gastroenterol J. 2014 Oct;2(5):383-90. doi: 10.1177/2050640614544315. PMID 25360316
- [Background] Inoue H, Ito H, Ikeda H, Sato C, Sato H, Phalanusitthepha C, Hayee B, Eleftheriadis N, Kudo SE. Anti-reflux mucosectomy for gastroesophageal reflux disease in the absence of hiatus hernia: a pilot study. Ann Gastroenterol. 2014;27(4):346-351. PMID 25330784
- [Background] Stefanidis D, Hope WW, Kohn GP, Reardon PR, Richardson WS, Fanelli RD; SAGES Guidelines Committee. Guidelines for surgical treatment of gastroesophageal reflux disease. Surg Endosc. 2010 Nov;24(11):2647-69. doi: 10.1007/s00464-010-1267-8. Epub 2010 Aug 20. No abstract available. PMID 20725747
- [Background] Gyawali CP, Fass R. Management of Gastroesophageal Reflux Disease. Gastroenterology. 2018 Jan;154(2):302-318. doi: 10.1053/j.gastro.2017.07.049. Epub 2017 Aug 5. PMID 28827081
- [Background] Huerta-Iga F, Tamayo-de la Cuesta JL, Noble-Lugo A, Hernandez-Guerrero A, Torres-Villalobos G, Ramos-de la Medina A, Pantoja-Millan JP; el Grupo Mexicano para el Estudio de la Enfermedad por Reflujo Gastroesofagico. [The Mexican consensus on gastroesophageal reflux disease. Part II]. Rev Gastroenterol Mex. 2013 Oct-Dec;78(4):231-9. doi: 10.1016/j.rgmx.2013.05.001. Epub 2013 Nov 28. Spanish. PMID 24290724